CLINICAL TRIAL: NCT03131999
Title: LAM Pilot Study With Imatinib Mesylate
Acronym: LAMP-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Charlie Strange, Professor of Pulmonary and Critical Care Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00044389
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2020-03-26 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Lymphangioleiomyomatosis
Keywords: VEGF-D; Imatinib mesylate; Sirolimus
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Imatinib Mesylate 400mg capsule (Experimental): 56 days of Imatinib mesylate 400 mg oral daily with or without co-administration of an mTOR inhibitor for 28 days. A dose reduction to 200 mg daily is allowed for toxicity.
  Interventions: Drug: Imatinib Mesylate 400Mg Capsule
- Placebo Capsule (Placebo Comparator): 56 days of Placebo with or without co-administration of an mTOR inhibitor for 28 days. A dose reduction is allowed for toxicity.
  Interventions: Drug: Placebo - Capsule

INTERVENTIONS:
Drug: Imatinib Mesylate 400Mg Capsule — Sirolimus or everolimus will be withdrawn after 28 days if used at baseline
  Other Names: Gleevec
  Arms: Imatinib Mesylate 400mg capsule
Drug: Placebo - Capsule — Sirolimus or everolimus will be withdrawn after 28 days if used at baseline
  Other Names: Placebo
  Arms: Placebo Capsule

SUMMARY:
This is a phase 1 clinical trial comparing imatinib mesylate to placebo for individuals with lymphangioleiomyomatosis (LAM).

DETAILED DESCRIPTION:
This is a double blind, adjusted parallel design, randomized clinical trial comparing imatinib mesylate 400 mg daily or matching placebo on the primary outcome of log transformed serum VEGF-D level in patients with LAM.

Sirolimus using patients will have co-administration of Imatinib mesylate or placebo for 28 days prior to sirolimus discontinuation.

The duration of 400 mg imatinib mesylate or placebo will be 56 days, a dose reduction is allowed for toxicity.

The primary endpoint will be the change in the log transformed VEGF-D one month after monotherapy imatinib mesylate or placebo.

Total trial duration is 2 months of drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Definite or Probable LAM
* FVC or Postbronchodilator FEV1 <90% predicted

Exclusion Criteria:

* Current or planned pregnancy or lactation
* Unwillingness to discontinue sirolimus
* Change in the dose or use of sirolimus within the past month
* Inability to perform spirometry
* Allergy or intolerance of albuterol and/or ipratropium
* Other serious illness that would impact the outcome of the study including cancer that has not received curative therapy, Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study), uncontrolled diabetes, chronic renal disease, chronic liver disease, or active uncontrolled infection
* Current lung transplant
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Current cigarette smoking
* Required use of warfarin, ketoconazole, itraconazole, clarithromycin, or rifampin during the 2 months of the study.
* Unwillingness to avoid grapefruit juice or St. Johns Wort during the study.
* Planned surgery during the 2 months of the study.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* Patient has received and other investigational agents within 28 days of first day of study drug dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Meinberg, Study Director — Congressionally Directed Medical Research Programs
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 Subjects signed consent, 2 subjects failed baseline evaluation and were not randomized. 1 subject was randomized, took 4 placebo pills and stopped (without side effects) and is deemed not evaluable.
Period: Overall Study
Arm/Group | Imatinib Mesylate 400mg Capsule | Placebo Capsule
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Withdrawal after 4 pills of placebo is not included in baseline population
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate 400mg Capsule | Placebo Capsule | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 50 (11) | 47.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Forced Expiratory Volume in 1 Second [Geometric Mean (Standard Deviation); unit: Percent predicted] | 59 (23.1) | 60 (15.4) | 59.5 (18.8)

OUTCOME MEASURES:

1. Primary Outcome: Serum VEGF-D
Description: Change in the square root of the intrasubject plasma VEGF-D
Time Frame: Before and 1 month after initiation of monotherapy imatinib mesylate or placebo
Measure: Mean (Standard Deviation); unit: Log transformed VEGF-D change pg/dL
Arm/Group | Imatinib Mesylate 400mg Capsule | Placebo Capsule
Number analyzed (Participants) | 8 | 7
Log transformed VEGF-D change pg/dL | 0.05 (0.10) | 0.07 (0.13)

2. Secondary Outcome: Adverse Events
Description: Adverse event and Serious Adverse Event numbers using the CTCAE Version 4.03 definitions
Time Frame: 3 months
Measure: Number; unit: number of events
Arm/Group | Imatinib Mesylate 400mg Capsule | Placebo Capsule
Number analyzed (Participants) | 8 | 7
number of events
  Adverse Events | 10 | 12
  Serious Adverse Events | 0 | 0

3. Other Pre Specified Outcome: Lung Function
Description: FEV1 % predicted change
Time Frame: 2 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: SGRQ
Description: Saint Georges Respiratory Questionnaire change
Time Frame: 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Imatinib Mesylate 400mg Capsule | Placebo Capsule
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 8/8 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate 400mg Capsule (N=8) | Placebo Capsule (N=7)
Nausea and/or vomitting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 3 (3) | 0 (0)
Insomnia (General disorders) | 0 | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Elevated Trough Sirolimus (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03131999/Prot_SAP_001.pdf